CLINICAL TRIAL: NCT01686542
Title: Circumferential Pulmonary Vein Isolation (CPVI) Plus Renal Sympathetic Modification Versus CPVI Alone for AF Ablation: a Pilot Study
Brief Title: CPVI Plus Renal Sympathetic Modification Versus CPVI Alone for AF（Atrial Fibrillation） Ablation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Director and Professor, Dept. of Cardiology, the second affiliated hospital of Chongqing Medical University, Chongqing Cardiac arrhythmias service center, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWAN-cpAF
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPVI+RSM group (Experimental): Circumferential pulmonary vein isolation (CPVI) plus renal sympathetic modification for atrial fibrillation ablation.
  Interventions: Procedure: CPVI plus renal sympathetic modification
- CPVI group (Active Comparator): Circumferential pulmonary vein isolation is done alone for atrial fibrillation.
  Interventions: Procedure: CPVI

INTERVENTIONS:
Procedure: CPVI plus renal sympathetic modification — CPVI plus renal denervation to reduce atrial arrhythmia recurrence.
  Other Names: Circumferential pulmonary vein isolation (CPVI); renal denervation; renal ablation
  Arms: CPVI+RSM group
Procedure: CPVI — CPVI alone to reduce atrial arrhythmia recurrence.
  Other Names: circumferential pulmonary vein ablation
  Arms: CPVI group

SUMMARY:
The study is designed as a randomized control trial. The purpose of this study is to observe the efficacy and safety of atrial fibrillation ablation, comparing circumferential pulmonary vein isolation (CPVI) plus renal sympathetic modification (RSM) with CPVI alone.

DETAILED DESCRIPTION:
Basic studies suggested that sympathetic nerves over-activity played an important role in the pathophysiological changes of arrhythmia occurrence. Present studies of renal ablation show a new method to decrease sympathetic nerves activity. Circumferential pulmonary vein isolation (CPVI) is an accepted ablation method for atrial fibrillation. The investigators plan to evaluate the efficiency and safety of CPVI plus renal sympathetic modification for atrial fibrillation ablation comparing with CPVI alone. The trial is going to recruit 100 patients randomized into two groups (CPVI+RSM group VS CPVI group = 50:50) with a follow-up duration of 4 years. The investigators aim to observe the relapse of atrial tachyarrhythmia lasting more than 30 seconds, the incidence of composite cardiovascular events after renal sympathetic modification, and safety and efficacy of the intervention, comparing with CPVI alone.

ELIGIBILITY:
Inclusion Criteria:

* • ≥ 18 years old, and ≤ 75 years old of age

  * more than half a year history of atrial fibrillation, no matter paroxysmal or persistent, with clinical symptom or ECG proved
  * be ineffective to at least one kind of anti-arrhythmic drugs treatment
  * echocardiography has done to except structural heart diseases such as congenital, valvular heart diseases and kinds of cardiomyopathy
  * estimated glomerular filtration rate (eGFR) of ≥ 45ml/min
  * is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

* • transesophageal echocardiography found thrombus in left atrial appendage

  * past history of atrial fibrillation surgical maze procedure
  * estimated glomerular filtration rate (eGFR) of < 45mL/min
  * has the history of renal restenosis or renal stents implantation
  * has experienced AMI（acute myocardial infarction） (old myocardial infarction is not excluded), unstable angina pectoris, cerebrovascular accidents, and alimentary tract hemorrhage within 3 months
  * patients with sick sinus syndrome
  * pregnant women
  * mental disorders
  * patients that have allergy to contrast agent
  * patients that do not go with follow-up
  * others such as researcher considers it is not appropriate to be included into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The relapse rate of atrial tachyarrhythmia | Four years
  Atrial tachyarrhythmia lasting more than 30 seconds consider relapsed

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China